CLINICAL TRIAL: NCT02486250
Title: Online Neuropsychological Test Validation Project With Imaging Pilot
Acronym: NVP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Johnson & Johnson (Industry); Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-12765
Record Dates: First submitted 2015-06-18; First posted 2015-07-01 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Validation of Online Cognitive Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

GROUPS / COHORTS (4):
- Main Study Recruits: Participants are recruited to come into a clinic and take supervised cognitive tests both online and paper/pencil as well as take unsupervised online cognitive tests at home. Participants will also be given a spit kit in clinic to determine ApOE Status.
  Interventions: Other: Validation Study
- MRI & PET Substudy: A subset of 34 participants from the Main Study Recruits will be invited to have an MRI and PET scan. The purpose of the sub-study is to obtain feasibility data for collecting longitudinal neuroimaging studies for participants in this sample.
  Interventions: Other: Validation Study
- ReVeRe 1: A subset of 250 participants from the Main Study Recruits and all MRI & PET Substudy participants will be invited to participate in ReVeRe 1. The purpose of ReVeRe is to validate an additional unsupervised online cognitive measure, administered via an iPad application.
  Interventions: Other: Validation Study
- ReVeRe 2: A subset of approximately 80 participants from the Main Study Recruits and MRI & PET Substudy participants will be invited to participate in ReVeRe 2. The purpose of ReVeRe 2 is to determine if performance on ReVeRe test battery is sensitive to amyloid positivity in cognitively intact older adults and also sensitive to longitudinal cognitive decline in this patient population.

INTERVENTIONS:
Other: Validation Study
  Groups: MRI & PET Substudy; Main Study Recruits; ReVeRe 1

SUMMARY:
This is a five year study conducted in cooperation with the Brain Health Registry (BHR), an internet-based registry which enrolls adult volunteers in order to facilitate clinical trials for the prevention of Alzheimer's disease (AD). The investigators goal is to validate the Brain Health Registry's online cognitive measures developed by Lumosity. Investigators will meet this goal by collecting data from the newly developed the BHR online cognitive screening battery along with standardized measures of memory, attention, executive functioning and speed of information processing currently used in clinical trials for Alzheimer's disease.

DETAILED DESCRIPTION:
This study is conducted in cooperation with the Brain Health Registry (BHR, CHR #12-09628), an internet-based registry which will enroll individuals in order to facilitate clinical trials for the prevention of Alzheimer's disease (AD) and other brain diseases and disorders.

The investigators goal is to validate the Brain Health Registry's online cognitive measures developed by Lumosity. Investigators will meet this goal by collecting data from the newly developed BHR online cognitive screening battery along with standardized measures of memory, attention, executive functioning and speed of information processing currently used in clinical trials for Alzheimer's disease.

Investigators will enroll 1000 subjects, 500 of whom will be recruited upon registering in the BHR. The other 500 subjects will be recruited from the Memory and Aging Center at the University of California, San Francisco (UCSF) and the Center for Imaging of Neurodegenerative Diseases (CIND) at the San Francisco VA Medical Center (SFVAMC). Demographic and clinical data will be obtained for each participant who will have 3 tests of cognitive function over a 2 week period: 1) unsupervised online cognitive testing, 2) supervised online cognitive testing, and 3) standard clinical neuropsychological assessments. The order in which cognitive evaluations are administered will be equally distributed within the sample so as to minimize practice effects. These subjects will also provide a saliva specimen in order to determine their ApoE genotype.

Additionally, investigators will also conduct a small pilot study of 34 subjects to obtain one 3 Tesla MRI scan and one PET scan in order to obtain feasibility data for collecting longitudinal neuroimaging studies for participants in this sample.

In addition to the main validation project and MRI/PET substudy, we will also run a substudy (n=330) that looks to validate an additional unsupervised online cognitive measure (administered via iPad application) called ReVeRe. ReVeRe, is an automated, self-administered measure of verbal memory (word list recall) that is modeled after the Rey Auditory Verbal Learning Test.

There are two substudies for ReVeRe:

ReVeRe 1 (n=250): This approximately 30 minute procedure will be administered initially during the NVP participant's clinic visit, and then will be collected remotely (by participants at home) on: (1) Day 7 after the initial clinic testing, (2) Day 21 after the initial clinic testing, and (3) ongoing at 6 month intervals through at least 18 months - for a total of 6 administrations.

ReVeRe 2 (n=80): This approximately 30 minute procedure will be administered initially 2 weeks after a follow up in-clinic visit, and then will be collected remotely in burst intervals. There will be three administrations at each time point (Day 0, 3, and 7), which will be collected every 6 months for 24 months after the in-clinic follow up visit. All participants in ReVeRe 2 will also receive an amyloid PET scan, as long as they did not already participate in the MRI/PET substudy.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 60 years and older
* Fluent in English
* Able to give informed consent
* Access and the ability to use the internet

Exclusion Criteria:

* Evidence or diagnosis of dementia
* Evidence of acute or uncontrolled medical illness
* Recent history (< 6 months) of abuse or dependence of drugs and/or alcohol
* Significant neurological disease (ex. Parkinson's disease, Epilepsy, Traumatic brain injury)

Additionally, subjects participating in the neuroimaging portion of the study, will be excluded for any of the following:

* Unable or unwilling to travel to SFVAMC and UCSF China Basin campuses for MRI and PET procedures
* Contraindications for MR exam, including claustrophobia, paramagnetic metal implants, inability to fit comfortably in MRI (BMI < 38)
* Clinically significant hepatic, renal, pulmonary, metabolic or endocrine disturbances as indicated by history which in the opinion of the Investigator might pose a potential safety risk to the subject
* Current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following:
* Cardiac surgery or myocardial infarction within the last 4 weeks
* Unstable angina
* Acute decompensated congestive heart failure or class IV heart failure
* Current significant cardiac arrhythmia or conduction disturbance, particularly those resulting in ventricular fibrillation, or causing syncope, or near syncope
* Uncontrolled high blood pressure
* QTc > 450 msec
* History of drug or alcohol abuse within the last year, or prior prolonged history of abuse
* Women of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception. Women of childbearing potential must not be pregnant or breastfeeding at screening.
* History of relevant severe drug allergy or hypersensitivity.
* Receiving an investigational medication under an FDA IND protocol within the last 30 days. Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication. Subjects who have ever participated in an experimental study with an amyloid targeting therapy (e.g., immunotherapy, secretase inhibitor) may not be enrolled without prior sponsor approval unless it can be demonstrated that the patient received only placebo in the course of the trial.
* Current clinically significant unstable medical comorbidities, as indicated by history that pose a potential safety risk to the subject
* Receiving a radiopharmaceutical for imaging or therapy within the past 24 hours prior to the imaging session for this study
* Opinion of the Investigator that the subject is otherwise an unsuitable for study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adults age 60 years and older
  * Fluent in English
  * Able to give informed consent
  * Access and the ability to use the internet
Sampling Method: Non-Probability Sample
Enrollment: 982 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Number of people recruited online for in-clinic study | 3 years
  Number of people recruited online for in-clinic study will help determine the feasibility of using the Brain Health Registry as a recruitment source for an in-clinic study at the SFVAMC.

SECONDARY OUTCOMES:
Difference between unsupervised cognitive test score vs. supervised cognitive test score | 3 years
  A primary goal of this study is to validate the unsupervised online cognitive screening battery with the supervised cognitive test score. We will meet this goal by collecting data from the newly developed BHR online cognitive screening battery along with standardized measures of memory, attention, executive functioning and speed of information processing currently used in clinical trials for Alzheimer's disease.

OTHER OUTCOMES:
Number of online recruited participants who successfully complete imaging component | 1 year
  Number of people recruited online for in-clinic study will help determine the feasibility of using the Brain Health Registry as a recruitment source for an amyloid PET imaging study.
Participants performance on ReVeRe test battery | 3 years
  The goal is to determine if the performance on the ReVeRe test battery is sensitive to amyloid positivity in cognitively intact older adults and is also sensitive to longitudinal cognitive decline in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weiner, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- BrainHealthRegistry.org, San Francisco, California, United States

REFERENCES:
- See also: This is the website for the Brain Health Registry. — http://www.brainhealthregistry.org